CLINICAL TRIAL: NCT05083169
Title: A Phase 3 Randomized Study Comparing Teclistamab in Combination With Daratumumab SC (Tec-Dara) Versus Daratumumab SC, Pomalidomide, and Dexamethasone (DPd) or Daratumumab SC, Bortezomib, and Dexamethasone (DVd) in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Teclistamab in Combination With Daratumumab Subcutaneously (SC) (Tec-Dara) Versus Daratumumab SC, Pomalidomide, and Dexamethasone (DPd) or Daratumumab SC, Bortezomib, and Dexamethasone (DVd) in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: MajesTEC-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109049; 64007957MMY3001 (Other: Janssen Research & Development, LLC); 2020-004742-11 (EudraCT Number); 2023-503441-55-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05463939 (Approved for marketing)
Record Dates: First submitted 2021-10-08; First posted 2021-10-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; pomalidomide; Dexamethasone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Teclistamab-daratumumab (Tec-Dara) (Experimental): Participants will receive teclistamab and daratumumab by subcutaneous (SC) injection. Step-up doses of teclistamab will be given prior to the first full dose.
  Interventions: Drug: Daratumumab; Drug: Teclistamab
- Arm B: DPd or DVd (Experimental): Participants will be randomized either to daratumumab, pomalidomide, dexamethasone (DPd) treatment to receive daratumumab SC injection; pomalidomide orally; dexamethasone orally or intravenously, or to Daratumumab, Bortezomib, Dexamethasone (DVd) treatment to receive daratumumab SC injection; bortezomib SC injection, and dexamethasone orally or intravenously.
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered SC injection.
Drug: Pomalidomide — Pomalidomide will be administered orally.
  Arms: Arm B: DPd or DVd
Drug: Dexamethasone — Dexamethasone will be administered orally or intravenously.
  Arms: Arm B: DPd or DVd
Drug: Bortezomib — Bortezomib will be administered SC injection.
  Arms: Arm B: DPd or DVd
Drug: Teclistamab — Teclistamab will be administered SC injection.
  Other Names: JNJ-64007957
  Arms: Arm A: Teclistamab-daratumumab (Tec-Dara)

SUMMARY:
The purpose of this study is to compare the efficacy of teclistamab daratumumab (Tec-Dara) with daratumumab subcutaneously (SC) in combination with pomalidomide and dexamethasone (DPd) or daratumumab SC in combination with bortezomib and dexamethasone (DVd).

ELIGIBILITY:
Inclusion Criteria:

* Documented multiple myeloma as defined by the criteria: a. multiple myeloma diagnosis according to the International Myeloma Working Group (IMWG) diagnostic criteria, b. measurable disease at screening as defined by any of the following: 1) serum M-protein level greater than or equal to (>=) 0.5 gram per deciliter (g/dL); or 2) urine M-protein level >=200 milligrams (mg)/24 hours; or 3) serum immunoglobulin free light chain >=10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Received 1 to 3 prior line(s) of antimyeloma therapy including a proteasome inhibitor (PI) and lenalidomide; a. participants who have received only 1 line of prior line of antimyeloma therapy must be lenalidomide refractory. Stable disease or progression on or within 60 days of the last dose of lenalidomide given as maintenance will meet this criterion
* Documented evidence of progressive disease based on investigator's determination of response by IMWG criteria on or after their last regimen
* Have an eastern cooperative oncology group (ECOG) performance status score of 0, 1, or 2 at screening and prior to the start of administration of study treatment
* Have clinical laboratory values within the specified range

Exclusion Criteria:

* Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug or its excipients. Additional exclusion criteria pertaining to specific study drugs include:

  1. A participant is not eligible to receive daratumumab subcutaneous (SC) in combination with pomalidomide and dexamethasone (DPd) as control therapy if any of the following are present: 1) Contraindications or life-threatening allergies, hypersensitivity, or intolerance to pomalidomide, 2) Disease that is considered refractory to pomalidomide per IMWG,
  2. A participant is not eligible to receive daratumumab SC in combination with bortezomib and dexamethasone (DVd) as control therapy if any of the following are present: 1) Contraindications or life-threatening allergies, hypersensitivity, or intolerance to bortezomib, 2) Grade 1 peripheral neuropathy with pain or Grade >= 2 peripheral neuropathy as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0, 3) Disease that is considered refractory to bortezomib per IMWG, 4) Received a strong cytochromes P450 (CYP3A4) inducer within 5 half-lives prior to randomization
* Received any prior B cell maturation antigen (BCMA)-directed therapy
* Has disease that is considered refractory to an anti-cluster of differentiation 38 (CD38) monoclonal antibody per IMWG
* Received a cumulative dose of corticosteroids equivalent to >=140 mg of prednisone within 14 days before randomization
* Received a live, attenuated vaccine within 4 weeks before randomization
* Plasma cell leukemia at the time of screening, Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes), or primary amyloid light chain amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2028-12-08 (Estimated); Study Completion 2028-12-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 5 years
  PFS is defined as the time from the date of randomization to the date of first documented disease progression, as defined in the International Myeloma Working Group (IMWG) criteria, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Response (Partial Response [PR] or Better) | Up to 5 years
  Overall response (PR or better) is defined as participants who have a PR or better per IMWG criteria.
Very Good Partial Response (VGPR) or Better | Up to 5 years
  VGPR or better is defined as participants who achieve a VGPR or better response per IMWG criteria.
Complete Response (CR) or Better | Up to 5 years
  CR or better is defined as participants who achieve a CR or better response per IMWG criteria.
Minimal Residual Disease (MRD)-negativity | Up to 5 years
  MRD-negativity is defined as participants who achieve MRD negativity at a threshold of 10^-5 at any timepoint after the date of randomization and before disease progression or start of subsequent antimyeloma therapy.
Progression Free Survival on Next-line Therapy (PFS2) | Up to 5 years
  PFS2 is defined as the time interval between the date of randomization and date of event, which is defined as progressive disease as assessed by investigator on the first subsequent line of antimyeloma therapy, or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 5 years
  OS is measured from the date of randomization to the date of the participant's death.
Time to Next Treatment (TTNT) | Up to 5 years
  TTNT is defined as the interval time from randomization to the start of subsequent antimyeloma treatment.
Duration of Response | Up to 5 years
  Duration of response will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease according to the IMWG response criteria, or death due to any cause, whichever occurs first.
Number of Participants with Adverse Events (AEs) by Severity | Up to 5 years
  Number of participants with AEs by Severity will be reported.
Serum Concentration of Teclistamab | Up to 5 years
  Serum samples will be analyzed to determine concentrations of teclistamab using a validated, specific, and sensitive method.
Number of Participants with Anti-drug Antibodies (ADAs) to Teclistamab and Daratumumab | Up to 5 years
  Number of participants with ADAs to teclistamab and daratumumab will be reported.
Time to Worsening of Symptoms | Up to 5 years
  Time to worsening is measured as the interval from the date of randomization to the start date of meaningful change.
Change from Baseline in Symptoms, Functioning, and Overall Health-related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC-QLQ-C30) | Baseline up to 5 years
  The EORTC-QLQ-C30 Version 3 includes 30 items in 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea/vomiting), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The responses are reported using a verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high/healthy level of functioning and a high score for the global health status represents high HRQoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Change from Baseline in Symptoms, Functioning, and Overall HRQoL as Assessed by Multiple Myeloma Symptom and Impact Questionnaire (MySIm-Q) Scale Score | Baseline up to 5 years
  The MySIm-Q is a disease-specific PRO assessment complementary to the EORTC-QLQ-C30. It includes 17 items resulting in a symptom subscale and an impact subscale. The recall period is the "past 7 days", and responses are reported on a 5-point verbal rating scale.
Change from Baseline in Symptoms, Functioning, and Overall HRQoL as Assessed by Patient-reported Outcomes Measurement Information System Short Form v2.0 - Physical Function 8c (PROMIS PF 8c) | Baseline up to 5 years
  The PROMIS-SD is used to assess self-reported perceptions of sleep quality, sleep depth and restoration associated with sleep. The 8-item short form will be used in this study, in which responses are scored 1 to 5 for each item. Higher overall score indicates more sleep disturbance.
Change from Baseline in Symptoms, Functioning, and Overall HRQoL as Assessed by Patient-reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE ) | Baseline up to 6 months
  The National Cancer Institute's (NCI's) PRO-CTCAE is an item library of common adverse events experienced by people with cancer that are appropriate for self-reporting of treatment tolerability. Each symptom selected for inclusion can be rated by up to 3 attributes characterizing the presence/frequency, severity, and/or interference of the AEs. It ranges from 0 to 4 with higher scores indicating higher frequency or greater severity/impact.
Change from Baseline in Symptoms, Functioning, and Overall HRQoL as Assessed by EuroQol Five Dimension Questionnaire 5-Level (EQ-5D-5L) | Baseline up to 5 years
  The EQ-5D-5L is a generic measure of health status. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Change from Baseline in Symptoms, Functioning, and Overall HRQoL as Assessed by Patient Global Impression - Severity (PGI-S) | Baseline up to 5 years
  The PGIS contains 2 questions on how the participant would currently rate severity of symptoms and impacts with a 7-day recall period. The response options are presented as a 5-point verbal rating scale from 1="none" to 5="very severe."
PFS in Participants with High-risk Molecular Features | Up to 5 years
  PFS in participants with high-risk molecular features will be reported.
Depth of Response in Participants in High-risk Molecular Features | Up to 5 years
  Depth of response in participants in high-risk molecular features will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (174):
- United States (18):
  - University of Alabama Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - Stanford University Medical Center, Stanford, California
  - Yale University, New Haven, Connecticut
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health System, Southfield, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Cancer Center, Memphis, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Argentina (3):
  - Hospital Aleman, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Privado Centro Medico de Cordoba, Córdoba
- Belgium (7):
  - ZAS Cadix, Antwerp
  - AZ St.-Jan Brugge-Oostende AV, Bruges
  - UZ Gent, Ghent
  - Hopital de Jolimont, Haine Saint Paul La Louviere
  - Az Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - Algemeen Ziekenhuis Delta, Roeselare
- Brazil (11):
  - Hospitais Integradaos da Gavea S/A - DF Star, Brasília
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina CEPEN, Florianópolis
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Hospital Sao Rafael, Salvador
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Hospital Paulistano, São Paulo
  - Clinica Medica Sao Germano S/S LTDA, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
- Canada (5):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency - Vancouver BC, Vancouver, British Columbia
  - QEII Health Sciences, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
- China (20):
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Third Xiangya Hospital of Central Sourth University, Changshashi
  - Beijing Chaoyang Hospital, Chaoyang District
  - West China Hospital Sichuan University, Chengdu
  - Fujian Meidical University Union Hospital, Fuzhou
  - Sun Yat -Sen University Cancer Center, Guangzhou
  - First affiliated Hospital of Zhejiang University, Hangzhou
  - Zhongda Hospital Southeast University, Nanjing
  - First Affiliated Hospital of Guangxi Medical University, Nanning
  - Shanghai Zhongshan Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Odense Universitets Hospital, Odense
  - Vejle Hospital, Vejle
- France (9):
  - CHU Henri Mondor, Créteil
  - CHRU de Lille Hopital Claude Huriez, Lille
  - CHU de Limoges Hopital Dupuytren, Limoges
  - C.H.U. Hotel Dieu - France, Nantes
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - CHU De Poitiers, Poitiers
  - Institut de Cancerologie Strasbourg Europe ICANS, Strasbourg
  - Pôle IUC Oncopole CHU, Toulouse
  - CHRU Hôpital Bretonneau, Tours
- Germany (10):
  - Universitätsklinikum Carl-Gustav-Carus Dresden, Dresden
  - Heinrich-Heine -Universitaet Duesseldorf, Düsseldorf
  - Evang. Krankenhaus Essen-Mitte gGmbH, Essen
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - St. Barbara-Klinik Hamm GmbH, Hamm
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Tuebingen, Tübingen
- Greece (3):
  - Alexandra General Hospital of Athens, Athens Attica
  - Anticancer Hospital of Thessaloniki Theageneio, Thessaloniki
  - G.Papanikolaou, Thessaloniki
- Italy (8):
  - U.O. Ematologia con Trapianto- AOU Policlinico di Bari, Bari
  - ASST Papa Giovanni XXIII Bergamo, Bergamo
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - IRCCS Policlinico San Matteo, Università degli studi di Pavi, Pavia
  - Università di Roma 'La Sapienza' - Ospedale Umberto 1°, Roma
  - A.O.U. Citta della Salute e della Scienza di Torino - Presidio Molinette, Turin
- Japan (19):
  - Fukuoka University Hospital, Fukuoka
  - Ogaki Municipal Hospital, Gifu
  - National Hospital Organization Mito Medical Center, Higashiibaraki-gun
  - Tokai University Hospital, Isehara
  - Shonan Kamakura General Hospital, Kamakura-shi
  - National Cancer Center Hospital East, Kashiwa
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Kumamoto University Hospital, Kumamoto
  - Kurume University Hospital, Kurume
  - National Hospital Organization Matsumoto Medical Center, Matsumoto
  - Nagoya City University Hospital, Nagoya
  - Hyogo Medical University Hospital, Nishinomiya Shi
  - National Hospital Organization Okayama Medical Center, Okayama
  - National Hospital Organization Hiroshima-Nishi Medical Center, Ōtake
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - National Hospital Organization Sendai Medical Center, Sendai
  - Japanese Red Cross Medical Center, Shibuya-ku
  - Iwate Medical University Hospital, Shiwa-gun
- Netherlands (5):
  - VU Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Sint Antonius Ziekenhuis - Afd.Interne - INT, Nieuwegein
  - Radboudumc, Nijmegen
  - Isala Kliniek, Zwolle
- Poland (7):
  - Klinika Hematologii i Transplantologii, UCK, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce
  - Centrum Onkologii Ziemi Lubelskiej im sw Jana z Dukli, Lublin
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
  - Specjalistyczny Szpital im dra Alfreda Sokolowskiego w Walbrzychu, Wałbrzych
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Russia (2):
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
- South Korea (7):
  - Kyungpook National University Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (15):
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. de Cabuenes, Gijón
  - Hosp. Univ. de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Son Espases, Palma
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
- Sweden (7):
  - Falu Lasarett, Falun
  - Sahlgrenska University Hospital, Gothenburg
  - Helsingborgs lasarett, Helsingborg
  - Sunderby Sjukhus, Luleå
  - Skanes universitetssjukhus, Lund
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Sjukhuset, Uppsala
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (4):
  - Ankara University Medical Faculty, Ankara
  - Ondokuz Mayis University, Atakum
  - Medipol University Hospital, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
- United Kingdom (6):
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Ninewells Hospital & Medical School, Dundee
  - Kings College Hospital, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Costa LJ, Bahlis NJ, Perrot A, Nooka AK, Lu J, Pawlyn C, Mina R, Caeiro G, Kentos A, Hungria V, Reece D, Niu T, Mylin AK, Hansen CT, Teipel R, Besemer B, Dimopoulos MA, Zamagni E, Yoshihara S, Kim K, Min CK, Geerts P, Van Leeuwen-Segarceanu E, Tyczynska A, Reguera JL, Johansson M, Hansson M, Turgut M, Grey M, Sidana S, Rodriguez-Otero P, Martinez-Lopez J, Hashmi H, Carson R, Kobos R, Sun W, Lantz K, Seifert A, Briseno-Toomey D, O'Rourke L, Rubin M, Vieyra D, Kang L, Mateos MV; MajesTEC-3 Trial Investigators. Teclistamab plus Daratumumab in Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2025 Dec 9. doi: 10.1056/NEJMoa2514663. Online ahead of print. PMID 41363801